CLINICAL TRIAL: NCT06780046
Title: Prospective Multicentric Cohort Study of Severe and Very Severe COPD Patients in Brazil.
Brief Title: Study That Will Evaluate the Brazilian Population With COPD.
Acronym: SCOPe
Status: Recruiting | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D5980R00117
Record Dates: First submitted 2025-01-13; First posted 2025-01-17 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: COPD (Chronic Obstructive Pulmonary Disease)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Observational, prospective, multicenter cohort study with consecutive inclusion of COPD patients. Eligible patients will be those with severe and very severe COPD according to the GOLD 2024 (Global Initiative for Chronic Obstructive Lung Disease) guidelines being followed at participating hospitals. The severity of COPD is related to the exacerbation rate, which in turn is related to the progression of the disease and the occurrence of complications and death. There is no national data on this subgroup.

DETAILED DESCRIPTION:
This is a prospective multicentre cohort, non-interventional study. The design is to have multiple medical centres representing the regions of Brazil. Each region has a different exposure to risk factors like tobacco smoke, biomass burning and environmental pollution, has a different population composition and density, degree of urbanization and education level. There are also some inferred genetic differences due to previous colonization and miscegenation. *CAT (COPD Assessment Test) OU CAAT (Chronic Airway Assesment Test) poderão ser usados intercambiavelmente. The patients will be enrolled in non-random consecutive method and will be followed up for 12 months.

There will be on-site visits at inclusion (V0), 6 and 12 months. There will tele-consults at 3 and 9 months to gather relevant clinical data, with special interest at exacerbation.

There will be 8 participating centres in Brazil, representing all 5 regions (North, Northeast, Midwest, Southeast and South). They will be Teaching Hospitals, Regional Reference Hospitals, Tertiary Hospitals or High Complexity Hospitals. The data will be collected on each site and will be adjudicated by the ARO Team.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes, aged 18 years or older, with confirmed COPD according to GOLD 2024: previous or current exposure and spirometry (FEV1/FVC =2 or CAT >=10); or
* GOLD E (>=2 moderate or 1 severe exacerbation - hospitalization); or
* GOLD 3 and 4 (FEV1 <50%).

Exclusion Criteria:

* Advanced fibrosing interstitial lung disease (extent >=50%); and/or
* High-risk pulmonary hypertension (on triple therapy); and/or
* Active cancer - on systemic therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults of both sexes with severe and very severe COPD being followed up at participating centers - referral hospitals distributed throughout the country. There are plans to include 693 patients from GOLD B, E, 3 and 4, who will be followed up for 12 months.
Sampling Method: Probability Sample
Enrollment: 693 (Estimated)
Dates: Start 2025-01-31 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of hospitalizations | through study completion, an average of 1 year
  Any need for hospitalization involving a hospital stay of more than 24 hours
Incidence of exacerbations | through study completion, an average of 1 year
  This is an acute event, with onset within 14 days, with increased symptoms: dyspnea, cough, expectoration
Incidence of Mortality | through study completion, an average of 1 year
  All deaths will be reviewed, determining the main cause of the fatal outcome.

SECONDARY OUTCOMES:
Incidence of vaccinated participants, with vaccines recommended by guidelines for patients with COPD | through study completion, an average of 1 year
  Vaccination rate for influenza, SARS-CoV-2, pneumococcus, adult double (or acellular triple bacterial) and triple viral.
Incidence of lung neoplasia | through study completion, an average of 1 year
  Results of any biopsies should be noted in the participant's medical record

CONTACTS AND LOCATIONS:
Locations (8):
- Brazil (8):
  - Research Site, Bahia
  - Research Site, Belém
  - Research Site, Brasília
  - Research Site, Campo Grande
  - Research Site, Florianópolis
  - Research Site, Santo André
  - Research Site, São Paulo
  - Research Site, Uberlândia

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/